CLINICAL TRIAL: NCT04393584
Title: Perioperative Chemotherapy With FOLFIRINOX Regimen or FLOT Regimen for Resectable Gastric or Esophagogastric Junction Adenocarcinoma (Type II-III): Open-label Randomized Phase 2/3 Trial
Brief Title: FOLFIRINOX vs FLOT Chemotherapy for Resectable Gastric or Esophagogastric Junction Adenocarcinoma
Acronym: RusGCG-01
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01
Record Dates: First submitted 2020-04-15; First posted 2020-05-19 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Stomach Neoplasms; Gastrointestinal Neoplasms; Docetaxel; Oxaliplatin; Fluoruracil; Irinotecan Hydrochloride
Keywords: gastric cancer; pathological complete; FLOT; FOLFIRINOX; gastrectomy; adenocarcinoma of the esophagogastric junction; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Neoplasms | interventions — Irinotecan; Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFIRINOX (Experimental): Irinotecan 180mg/m2 d1, d1-2 5-FU 2450 mg/m², d1 Leucovorin 200 mg/m², d1 Oxaliplatin 85 mg/m², d1 every two weeks (q2w) 4 cycles (4-8 weeks) pre-OP and 4 cycles (6-12 weeks) post-OP
  Interventions: Drug: Irinotecan; Drug: 5-FU; Drug: Leucovorin; Drug: Oxaliplatin
- FLOT (Active Comparator): d1 Docetaxel 50mg/m2, d1-2 5-FU 2600 mg/m², d1 Leucovorin 200 mg/m², d1 Oxaliplatin 85 mg/m² every two weeks (q2w) 4 cycles (4-8 weeks) pre-OP and 4 cycles (6-12 weeks) post-OP
  Interventions: Drug: 5-FU; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Irinotecan — d1 Irinotecan 180mg/m² every two weeks
  Arms: FOLFIRINOX
Drug: 5-FU — d1-2 5-FU 2450 mg/m² every two weeks
Drug: Leucovorin — d1 Leucovorin 200 mg/m² every two weeks
Drug: Oxaliplatin — d1 Oxaliplatin 85 mg/m² every two weeks
Drug: Docetaxel — d1 Docetaxel 50mg/m2 every two weeks
  Arms: FLOT

SUMMARY:
Patients with resectable adenocarcinoma of the stomach or the esophagogastric junction (II-III type by Siewert) without previous therapy will be treated with one of two chemotherapy combinations before and after surgery. One half of the patients gets 5-Fluorouracil (5-FU), Leucovorin, Oxaliplatin and Docetaxel (FLOT), the others 5-Fluorouracil (5-FU), Leucovorin, Oxaliplatin and Irinotecan (FOLFIRINOX). Main objective of the study is median overall survival.

DETAILED DESCRIPTION:
538 Patients with resectable (cT4cN0 or cT1-4 and cN+, cM0) adenocarcinoma of the stomach or the esophagogastric junction without previous therapy will be included in this study. After randomization patients receive perioperatively 4 cycles FLOT or FOLFIRINOX, followed by a restaging of the tumour status and surgery. Subsequently another 4 cycles of FLOT or FOLFIRNOX are applicated.

ELIGIBILITY:
Inclusion Criteria:

1. сT4 cN0 or cT1-4 cN+ histologically proven adenocarcinoma of the esophagogastric junction (Siewert type II-III) or the stomach without distant metastases (M0)
2. No previous cytostatic chemotherapy or radiation therapy
3. Age 18-70 years (female and male)
4. Eastern Cooperative Oncology Group ≤ 2
5. Surgical resectability
6. Neutrophils> 2.000/µl
7. Platelets > 100.000/µl
8. Normal value of Serum Creatinin
9. Albumin level > 29 г/л
10. Aspartate transaminase (AST) or alanine transaminase (ALT) less than 3 times the upper limits of normal (ULN)
11. Total Bilirubin less than 1.5 times the ULN
12. Written informed consent.

Exclusion Criteria:

1. Previous cytostatic chemotherapy or radiation therapy
2. Distant metastases or all primarily not resectable stages
3. Cancer relapse
4. Complicated gastric cancer (perforation, bleeding, sub or decompensated stenosis, dysphagia IV)
5. Diarrhea ≥ 2 according to the criteria of Common Terminology Criteria for Adverse Events (CTCAE) version 4.1;
6. Hypersensitivity against 5- Fluorouracil, Leucovorin, Oxaliplatin, Epirubicin and Docetaxel
7. Existence of contraindications against 5- Fluorouracil, Leucovorin, Oxaliplatin, Irinotecan or Docetaxel
8. Active coronary heart disease, Cardiomyopathy or cardiac insufficiency stage III-IV according to New York Heart Association (NYHA)
9. Severe non-surgical accompanying disease or acute infection (uncontrolled arterial hypertension, diabetes mellitus, stroke less than 6 months old, mental disorders, other tumors and others)
10. Malignant secondary disease, dated back < 5 years (exception: In-situ-carcinoma of the cervix uteri, adequately treated skin basal cell carcinoma)
11. Peripheral polyneuropathy > Grad II
12. Liver dysfunction (AST)/ALT>3,0xULN, ALT>3xULN, Bilirubin>1,5xULN)
13. Serum Creatinin >1,0xULN
14. Chronic inflammable gastro-intestinal disease
15. Inclusion in another clinical trial
16. Pregnancy or lactation
17. Hepatitis B or C in the active stage
18. Human immunodeficiency virus(HIV) infected
19. Serious concomitant somatic and mental illnesses / deviations or territorial causes that may prevent the patient from participating in the protocol and observing the protocol schedule
20. Foreigners or persons with limited legal status

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 538 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
median overall survival | 2 years

SECONDARY OUTCOMES:
Pathologic complete response rate | 1 month after surgery
Disease free survival | 2 years
Perioperative Morbidity and Mortality | 1 months after surgery
R0-Resection rate | 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Stilidi, PhD, Principal Investigator — NN Blokhin National Medical Research Center of Oncology
Locations (1):
- Aleksei Kalinin, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No